CLINICAL TRIAL: NCT05429996
Title: Decrypting the Ultrastructural Collagen Markers Using Quantitative Nano Histology: A Quest for Newer Diagnostic Test in Hypermobile Ehlers-Danlos Syndrome
Brief Title: Ultrastructural Collagen Markers in Ehlers Danlos Syndromes
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Nimish Mittal, Staff Physician/Clinical Investigator, University Health Network, Toronto
Other Study IDs: 21-5542.0
Record Dates: First submitted 2022-06-17; First posted 2022-06-24 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Ehlers-Danlos Syndrome; Classical Ehlers-Danlos Syndrome; Hypermobile EDS (hEDS)
MeSH Terms: conditions — Ehlers-Danlos Syndrome; Ehlers-Danlos syndrome type 1; Ehlers-Danlos syndrome type 3

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Skin biopsy samples of individual with cEDS and hEDS will be collected for the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with hypermobile EDS: Skin biopsy collection
  Interventions: Other: Skin Biopsy
- Individuals with classical EDS: Skin biopsy collection
  Interventions: Other: Skin Biopsy

INTERVENTIONS:
Other: Skin Biopsy — Skin biopsy specimens will be collected for both groups and subjected to quantitative nano histology using atomic force microscopy to assess for structural profile of a single collagen fibril

SUMMARY:
Establishing the diagnosis of Ehlers Danlos Syndromes (EDS)/generalized hypermobility spectrum disorders (G-HSD) is often problematic for patients. The absence of a precise unifying diagnosis in patients results in a significant emotional burden on the patient and caregivers, not to mention the hidden costs, including multiple recurring visits to several medical specialists and associated social and economic costs. To date, while collagen ultra-scale morphological heterogeneity has been used to comment on an EDS diagnosis, the mechanical properties of the collagen remain mostly unexplored.

From a biophysical point of view, collagen affected with hEDS can be described as biomechanically deficient. In the case of EDS, the skin's abnormal elasticity can be directly related to the organization of the collagen network within the dermis. Quantitative Nanohistology (QNH) is a newer method to evaluate both the structural and mechanical properties of collagen in-situ histological sections.

Therefore, the aim of this study is to define histo-biophysical markers of two most common types of EDS i.e. classical EDS (cEDS) & hypermobile EDS (hEDS) at the single collagen fibrils level and matrix and to further explore the origin of collagen fibril properties deficiency in hEDS and cEDS.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 60 years who can provide informed consent in English
* Able to read, speak, and comprehend English without the assistance of a translator
* Have been diagnosed with hypermobile EDS as per the 2017 EDS criteria; or with genetically confirmed classical EDS (age and sex-matched). This diagnosis is carried out by the UHN GoodHope EDS clinic routinely for all patients on the basis of clinical exam and genetic testing, if indicated.

Exclusion Criteria:

* Subjects under the age of 18
* Unable to speak, read and comprehend English
* Unable to provide consent (cognitive impairment)
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with classical EDS and hypermobile EDS
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-10-31 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
to analyze percentage prevalence of abnormal morphological markers of single collagen fibril using atomic force microscopy | 3 months
  systemic nanoscale imaging to investigate the presence of morphological markers associated with each EDS type and compared to the normative data from the Bozec-lab obtained from healthy volunteers. These markers include fibrils D-banding periodicity, unwinding of the fibrils, variation in fibrils registration, and finally, cylindrical homogeneity (of the fibril

CONTACTS AND LOCATIONS:
Locations (1):
- GoodHope EDS - Toronto General Hospital, Toronto, Ontario, Canada